CLINICAL TRIAL: NCT01787318
Title: Effect of the Insupatch on Automated Closed-loop Glucose Control in Type 1 Diabetes
Acronym: IPCL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIC # 1208010682
Record Dates: First submitted 2013-01-16; First posted 2013-02-08 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ePID closed loop system using Insupatch (Experimental): Insupatch activated at mealtimes
  Interventions: Device: ePID closed loop system; Device: InsuPatch
- ePID closed loop system without InsuPatch (Active Comparator): InsuPatch will not be activated at mealtimes
  Interventions: Device: ePID closed loop system

INTERVENTIONS:
Device: ePID closed loop system — Insulin pump controlled by closed loop unit and algorithm
Device: InsuPatch — device which applies local heating at 40 degrees Celsius to the vicinity of the subcutaneous insulin infusion insertion site
  Arms: ePID closed loop system using Insupatch

SUMMARY:
This research study designed to look at how well adolescents' and young adults' blood sugars can be controlled with a "closed loop artificial pancreas" using a continuous glucose sensor, an insulin pump, and a computer program that automatically determines how much insulin to give based on the glucose level. The investigators will also study the effect of wearing a small heating patch, the InsuPatch, at the site of insulin infusion, on the ability of the closed loop system to control the blood sugar levels and to reduce the rise in glucose levels after meals.

DETAILED DESCRIPTION:
This is an open-label, single-center, randomized crossover study evaluating the performance of a closed-loop (CL) insulin delivery system using a subcutaneous glucose sensor and an external insulin pump comparing the peak post-prandial glucose levels and the post-prandial glucose AUC during either CL control alone or CL control with the InsuPatch in an inpatient hospital research unit (HRU) setting. The closed loop visit consists of approximately 67 hours over 4 days and 3 nights.

ELIGIBILITY:
Inclusion Criteria:

1. age 12-40 years
2. clinical diagnosis of type 1 diabetes
3. duration of type 1 diabetes ≥ 1 year
4. HbA1c ≤ 9 %
5. Treated with pump therapy for at least 3 months
6. Body weight > 40 kg

Exclusion Criteria:

1. Insulin resistant (defined as requiring > 1.5 units/kg/day at time of study enrollment
2. Presence of any medical or psychiatric disorder that may interfere with subject safety or study conduct
3. Use of any medications (besides insulin) known to blood glucose levels, including oral or other systemic glucocorticoid therapy. Inhaled, intranasal, or rectal corticosteroid use is allowed along as not given within 4 weeks of admission. Use of topical glucocorticoids is allowable as long as affected skin area does not overlap with study device sites. Subjects using herbal supplements will be excluded, due to the unknown effects of these supplements on glucose control
4. History of poor wound healing, heat sensitivity, or diminished skin integrity.
5. History of hypoglycemic seizure within last 3 months
6. Anemic (low hematocrit), or evidence of renal insufficiency (elevated serum creatinine)
7. Female subjects who are pregnant, lactating, or unwilling to be tested for pregnancy
8. Subjects unable to give consent / permission / assent

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Peak Post-Prandial Glucose Excursions | 48 hours
  Peak post-prandial plasma glucose excursions after breakfast, lunch, and dinner on days #2 and #3. One day with InsuPatch activated and one day without InsuPatch activated

SECONDARY OUTCOMES:
Total Area Under Curve of the meal-related glucose excursion over target | 48 hours
Nadir glucose levels following the meals | 48 hours
Mean 24 hour glucose levels | 48 hours
Mean daytime and nighttime glucose levels | 48 hours
Peak post-prandial insulin levels following meals | 48 hours
Area Under Curve meal-related insulin excursion following meals | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Weinzimer, MD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States